CLINICAL TRIAL: NCT02845752
Title: A Randomized, Crossover, Placebo Controlled, Double-blind Trial of the Effect of STIOLTO™ RESPIMAT® on Central and Peripheral Components of Fatigue During Exercise in Chronic Obstructive Pulmonary Disease
Brief Title: The Effect of STIOLTO™ RESPIMAT® on Fatigue in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Richard Casaburi, Professor, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1237.55; 21394-01 (Other: Los Angeles Biomedical Research Institute)
Record Dates: First submitted 2016-07-24; First posted 2016-07-27 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol; Tiotropium Bromide; olodaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stiolto Respimat (Active Comparator): Two actuations of Stiolto Respimat inhaler, taken once daily for 7 days. After a washout period of 14 days, participants will then receive matching Placebo for 7 days.
  Interventions: Drug: Stiolto Respimat; Drug: Placebo Respimat
- Placebo Respimat (Placebo Comparator): Two actuations of Placebo Respimat inhaler, taken once daily for 7 days. After a washout period of 14 days, participants will then receive matching Placebo for 7 days.
  Interventions: Drug: Stiolto Respimat; Drug: Placebo Respimat

INTERVENTIONS:
Drug: Stiolto Respimat — Oral inhalation spray
  Other Names: Tiotropium Bromide and Olodaterol
Drug: Placebo Respimat — Oral inhalation spray

SUMMARY:
The purpose of this study is to determine whether exercise can be prolonged in COPD can by the inhaled bronchodilator Stiolto Respimat. The study will identify whether any endurance benefit is due to reduction in fatigue that originates within the skeletal muscles and/or from effects on neural activation of the skeletal muscles.

DETAILED DESCRIPTION:
Patients with chronic obstructive pulmonary disease (COPD) have reduced exercise tolerance. One mechanism for this is thought to be due to dynamic hyperinflation during exercise (an increase in the end-expiratory lung volume) that contributes to the sensation of breathlessness. Whether this also contributes to inhibiting motor recruitment, and reduces the available power output (termed performance fatigue; PF), is not well understood. Preliminary data suggests that many COPD patients, unlike healthy subjects, stop exercise with a 'skeletal muscle power reserve' i.e. the ability to acutely increase muscle power output. This suggests that they are limited in the exercise task by mechanisms other than acute intramuscular limitations to power production (termed muscle fatigue; MF). Exercise tolerance is increased by treatment with the fixed-dose combination bronchodilator, STIOLTO™ RESPIMAT®. We hypothesize that increased exercise tolerance with STIOLTO™ RESPIMAT® (reduced performance fatigue; PF) will be mediated by a combination of: 1) reduced inhibition of muscle activation (termed activation fatigue; AF) allowing patients to drive their leg muscles harder, and thus; 2) increased muscle fatigue (MF).

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following criteria: (a) Patients must be in a stable state of their disease with no exacerbation within the previous 4 weeks; and (b) At visit 1 spirometric must demonstrate a post-bronchodilator FEV1 <80% of predicted normal and a post-bronchodilator FEV1/FVC <70%.
* At visit 1, patients will demonstrate appreciable reversibility, defined as a 12% increase in FEV1 in response to albuterol administration.
* Baseline dyspnea index focal score ≤ 9.
* Male or female patients, between 45 and 90 years (inclusive) of age.
* Patients must be current or ex-smokers with a smoking history of more than 10 pack-years
* Patients must be able to perform technically acceptable pulmonary function tests must be able to complete multiple symptom-limited cycle ergometry tests.
* Patients must be able to inhale medication in a competent manner from the inhalers used in the study.

Exclusion Criteria:

* Patients with a significant disease other than COPD; a significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the study, (ii) influence the results of the study, or (iii) cause concern regarding the patient's ability to participate in the study.
* Patients with a documented history of asthma. For patients with allergic rhinitis or atopy, medical records will be required to verify that the patient does not have asthma.
* Patients with any of the following conditions:

  1. A history of myocardial infarction within 1 year of screening visit.
  2. Unstable or life-threatening cardiac arrhythmia.
  3. Hospitalized for heart failure within the past year.
  4. Known active tuberculosis.
  5. A malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last two years (patients with treated basal cell carcinoma are allowed).
  6. A history of life-threatening pulmonary obstruction within the past two years.
  7. A history of cystic fibrosis.
  8. Clinically evident bronchiectasis.
  9. A history of significant alcohol or drug abuse within the past two years.
  10. Any contraindications for exercise testing as outlined below (see contraindications to exercise).
  11. Patients who have undergone thoracotomy with pulmonary resection.
* Patients being treated with oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
* Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during clinic visits.
* Patients who desaturate to SpO2 <85% on screening incremental exercise testing.
* Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit or patients who are currently in a pulmonary rehabilitation program.
* Patients who have a limitation of exercise performance as a result of factors other than fatigue or exertional dyspnea, such as arthritis in the leg, angina pectoris or claudication or morbid obesity.
* Patients with a constant power cycle ergometry endurance time less than 4 or greater than 10 minutes after work rate adjustment procedures (described below).
* Patients who have taken an investigational drug within one month or six half-lives (whichever is greater) prior to screening visit (Visit 1).
* Pregnant or nursing women.
* Women of childbearing who have the potential not to be using a highly effective method of birth control. Female patients will be considered to be of childbearing potential unless surgically sterilized by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years.
* Patients who are currently participating in another interventional study.
* Patients who are unable to comply with pulmonary medication restrictions prior to randomization.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Casaburi, PhD, MD, Principal Investigator — LABioMed at Harbor-UCLA Medical Center; Harry Rossiter, PhD, Principal Investigator — LABioMed at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao M, Calmelat RA, Kierstead P, Carraro N, Stringer WW, Porszasz J, Casaburi R, Rossiter HB. A randomized, crossover, placebo controlled, double-blind trial of the effects of tiotropium-olodaterol on neuromuscular performance during exercise in COPD. J Appl Physiol (1985). 2022 May 1;132(5):1145-1153. doi: 10.1152/japplphysiol.00332.2021. Epub 2022 Mar 24. PMID 35323052

RESULTS

PARTICIPANT FLOW:
Groups:
- Stiolto Respimat, Then Placebo Respimat: Participants first received Stiolto Respimat inhaler (two actuations, once daily for 7 days). After a washout period of 14 days, participants will then received Placebo Respimat inhaler (two actuations, once daily for 7 days).
- Placebo Respimat, Then Stiolto Respimat: Participants first received Placebo Respimat inhaler (two actuations, once daily for 7 days). After a washout period of 14 days, participants will then received Stiolto Respimat inhaler (two actuations, once daily for 7 days).
Period: First Intervention (7 Days)
Arm/Group | Stiolto Respimat, Then Placebo Respimat | Placebo Respimat, Then Stiolto Respimat
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | Stiolto Respimat, Then Placebo Respimat | Placebo Respimat, Then Stiolto Respimat
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Stiolto Respimat, Then Placebo Respimat | Placebo Respimat, Then Stiolto Respimat
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stiolto Respimat, Then Placebo Respimat | Placebo Respimat, Then Stiolto Respimat | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 63 [58 to 64] | 71 [53 to 73] | 64 [58 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: The Magnitude of Change in Isokinetic Power (Performance Fatigue, PF) Associated With Stiolto Respimat Compared With Placebo Respimat at Isotime During Constant Work Rate Exercise (CWR)
Description: Constant work rate (CWR) exercise causes fatigue. Fatigue is measured by the difference between pre-CWR and post-CWR maximal voluntary isokinetic power i.e. how much maximal voluntary isokinetic power declines during CWR. The magnitude of fatigue is measured in watts at the time of the shortest exercise duration in either study arm, which is termed "isotime". A smaller value (in watts) of performance fatigue means that the intervention was associated with less fatigue after a given CWR exercise duration (i.e. at isotime).
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: watts
Groups:
- Stiolto Respimat: Stiolto Respimat inhaler (two actuations, taken once daily for 7 days).
- Placebo Respimat: Placebo Respimat inhaler (two actuations, taken once daily for 7 days).
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
watts | 75 [53 to 103] | 77 [61 to 117]

2. Secondary Outcome: The Magnitude of Change Electromyographic (EMG) Muscle Activity (Activation Fatigue, AF) Associated With Stiolto Respimat Compared With Placebo Respimat at Isotime During Constant Work Rate Exercise (CWR)
Description: Constant work rate (CWR) exercise causes fatigue and reduces muscle activation. The relationship between muscle activation and power is measured at baseline (unfatigued condition). Fatigue is measured by the difference between pre-CWR and post-CWR maximal voluntary isokinetic power i.e. how much maximal voluntary isokinetic power declines during CWR. The fraction of fatigue that is ascribed to reduced muscle activity is then calculated. The magnitude of activation fatigue is measured in EMG activity and expressed in watts at the time of the shortest exercise duration in either study arm, which is termed "isotime". A smaller value (in watts) of activation fatigue means that the intervention was associated with a less reduction in EMG activity after a given CWR exercise duration (i.e. at isotime).
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: watts
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
watts | 58 [33 to 74] | 50 [27 to 80]

3. Secondary Outcome: Exercise Endurance Time During CWR Cycling Exercise
Description: The duration in seconds for which constant work rate (CWR) cycling exercise could be tolerated prior to voluntary termination of exercise.
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
seconds | 297 [253 to 352] | 274 [222 to 326]

4. Secondary Outcome: Change From Period Baseline in the Exercise-isotime Inspiratory Reserve Volume During CWR
Description: Inspiratory reserve volume (IRV) measured during CWR cycling exercise at the time of the shortest duration of each intervention arm (isotime). A greater IRV would reflect a beneficial response to intervention.
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: Liters
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
Liters | 0.54 [0.26 to 0.86] | 0.46 [0.31 to 0.60]

5. Secondary Outcome: Change From Period Baseline in the Exercise-isotime Inspiratory Capacity During CWR
Description: Inspiratory capacity (IC) measured during constant work rate (CWR) cycling exercise at the time of the shortest duration of each intervention arm (isotime). A greater IC would reflect a beneficial response to the intervention.
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: Liters
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
Liters | 1.91 [1.64 to 2.48] | 1.88 [1.71 to 2.25]

6. Secondary Outcome: Change From Period Baseline in the Forced Expiratory Volume in 1 Second (FEV1)
Description: This outcome describes the the effect of the intervention on forced expiratory volume in 1 second (FEV1) during resting spirometry. A greater FEV1 would reflect a positive benefit of the intervention.
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: Liters
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
Liters | 1.81 [1.58 to 1.98] | 1.72 [1.29 to 1.99]

7. Secondary Outcome: Change From Period Baseline in the Exercise-isotime in Pulse Oximeter Oxygen Saturation During CWR
Description: Percentage of arterial hemoglobin that is saturated with oxygen, measured using pulse oximetry during constant work rate (CWR) cycling exercise at the time of the shortest duration of each intervention arm (isotime). A greater pulse oximeter oxygen saturation would reflect a beneficial response to the intervention.
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: percent of hemoglobin saturated with O2
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
percent of hemoglobin saturated with O2 | 99.0 [97.3 to 100.0] | 98.5 [97.8 to 100.0]

8. Secondary Outcome: Change From Period Baseline in the Exercise-isotime Ventilation During CWR
Description: Minute ventilation (VE) measured during constant work rate (CWR) cycling exercise at the time of the shortest duration of each intervention arm (isotime). A lesser VE would reflect a beneficial response to the intervention.
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: Liters/minute
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
Liters/minute | 50.20 [44.65 to 55.45] | 45.25 [42.95 to 55.43]

9. Secondary Outcome: Change From Period Baseline in the Exercise-isotime Oxygen Uptake (VO2) During CWR
Description: Pulmonary oxygen uptake (VO2) measured during constant work rate (CWR) cycling exercise at the time of the shortest duration of each intervention arm (isotime). A lesser VO2 would reflect a beneficial response to the intervention.
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: Liters/minute
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
Liters/minute | 1.279 [0.996 to 1.462] | 1.219 [1.070 to 1.452]

10. Secondary Outcome: Change From Period Baseline in the Exercise-isotime Frontal Lobe Oxygen Saturation During CWR
Description: Tissue saturation of hemoglobin with oxygen is measured by spatially resolved near-infrared spectroscopy from the frontal lobe during constant work rate (CWR) cycling exercise at the time of the shortest duration of each intervention arm (isotime). A greater frontal lobe oxygen saturation at isotime would reflect a beneficial response to the intervention.
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: Percent of hemoglobin saturated with O2
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
Percent of hemoglobin saturated with O2 | 62.5 [58.0 to 67.0] | 62.8 [56.6 to 65.9]

11. Secondary Outcome: Change From Period Baseline in the Exercise-isotime Muscle Oxygen Saturation During CWR
Description: Tissue saturation of hemoglobin plus myoglobin with oxygen is measured by spatially resolved near-infrared spectroscopy from the vastus lateralis muscle during constant work rate (CWR) cycling exercise at the time of the shortest duration of each intervention arm (isotime). A greater muscle oxygen saturation at isotime would reflect a beneficial response to the intervention.
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: % of O2 saturated hemoglobin+myoglobin
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
% of O2 saturated hemoglobin+myoglobin | 54.5 [43.9 to 60.8] | 53.4 [44.2 to 58.7]

12. Secondary Outcome: Change From Period Baseline in the Exercise-isotime Borg CR-10 Rating of Perceived Dyspnea During CWR
Description: Borg rating of perceived shortness of breath (dyspnea) were measured on a category-ratio scale from 0 to 10 (CR-10) during constant work rate (CWR) cycling exercise at the time of the shortest duration of each intervention arm (isotime). A lower CR-10 score for dyspnea at isotime would reflect a beneficial response to the intervention.
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
scores on a scale | 3 [2 to 4] | 2.5 [1 to 4]

13. Secondary Outcome: Change From Period Baseline in the Exercise-isotime Borg CR-10 Rating of Perceived Leg Fatigue During CWR
Description: Borg rating of perceived tiredness on the legs (leg fatigue) were measured on a category-ratio scale from 0 to 10 (CR-10) during constant work rate (CWR) cycling exercise at the time of the shortest duration of each intervention arm (isotime). A lower CR-10 score for leg fatigue at isotime would reflect a beneficial response to the intervention.
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
scores on a scale | 3 [2 to 4] | 2.5 [1 to 4]

14. Secondary Outcome: Change From Period Baseline in the Pre/Post Exercise-induced Decline in Peak Isokinetic Power Normalized to the Measured Muscle Activity (Muscle Fatigue, MF) During CWR
Description: Constant work rate (CWR) exercise causes muscle fatigue (MF) and reduces muscle activation (activation fatigue; AF). The relationship between muscle activity (using EMG) and power is measured at baseline (unfatigued condition). Fatigue is measured by the difference between pre-CWR and post-CWR maximal voluntary isokinetic power i.e. how much maximal voluntary isokinetic power declines during CWR. The fraction of the total fall in voluntary isokinetic power (total fatigue) that is ascribed to reduced muscle activity is then calculated from the reduction in EMG activity. The remainder is ascribed to muscle fatigue (MF) and expressed as a percentage of total fatigue. This measurement was made at peak exercise. A smaller value (%) of MF would be associated with a beneficial response to the intervention.
Time Frame: Baseline and day 7 of each treatment period
Measure: Median (Inter-Quartile Range); unit: percentage of total fatigue
Arm/Group | Stiolto Respimat | Placebo Respimat
Number analyzed (Participants) | 14 | 14
percentage of total fatigue | 20.9 [0 to 51.9] | 25.4 [14.0 to 68.41]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Stiolto Respimat | Placebo Respimat
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT02845752/Prot_SAP_000.pdf